CLINICAL TRIAL: NCT00248534
Title: A Phase II Study of Rituximab and Temozolomide in Recurrent Primary CNS Lymphoma
Brief Title: Rituximab, Temozolomide, and Methylprednisolone in Treating Patients With Recurrent Primary CNS Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual/lack of resources/low priority due to combining 2 consortia
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTC05-01; NABTC-05-01; CDR0000445289 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02673 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U01CA062399 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Methylprednisolone; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV Rituximab (Experimental): IV Rituximab 750mg/m2 single infusion every week for up to 4 weeks.
  Induction: Rituximab (750mg/m2) Day 1, 8, 15 and 22 and Temozolomide [TMZ] (150mg/m2) days 1-7 and 15-21, followed by six cycles of consolidation TMZ 150-200mg/m2 x5/28days, followed by maintenance with methylprednisolone (1g IV every 28days) until progression
  Interventions: Biological: rituximab; Drug: methylprednisolone; Drug: temozolomide

INTERVENTIONS:
Biological: rituximab — given IV days 1,8, 15 and 22
Drug: methylprednisolone — 2hr IV every 28 days post consolidation cycles of Temozolomide (TMZ) (6 cycles TMZ = Consolidation cycles)
Drug: temozolomide — Induction Days 1-7 and 15-21 (150mg/m2 PO) Consolidation days 1-5 every 28 days X 6 cycles
  Other Names: TMZ

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as temozolomide and methylprednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Rituximab may help chemotherapy kill more cancer cells by making cancer cells more sensitive to the drugs. Giving rituximab together with temozolomide and methylprednisolone may be an effective treatment for primary CNS non-Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well giving rituximab together with temozolomide and methylprednisolone works in treating patients with recurrent primary CNS non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with recurrent primary CNS non-Hodgkin's lymphoma treated with rituximab, temozolomide, and methylprednisolone.

Secondary

* Determine the overall and 6-month progression-free survival of patients treated with this regimen.

OUTLINE: Induction therapy: Patients receive rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 and oral temozolomide daily on days 1-7 and 15-21. After day 28, patients with stable disease or better proceed to consolidation therapy.

Consolidation therapy: Patients receive oral temozolomide daily on days 1-5. Treatment repeats every 28 days for up to 6 courses. Patients achieving a complete remission proceed to maintenance therapy.

Maintenance therapy: Patients receive methylprednisolone IV over 2 hours on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within approximately 13.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS non-Hodgkin's lymphoma by brain biopsy, positive cerebrospinal fluid cytology, or vitrectomy

  * Recurrent disease
* Measurable disease, define as bi-dimensionally measurable lesions with clearly defined margins by brain MRI or CT scan

  * Radiographical evidence of tumor progression by MRI or CT scan
  * Steroid therapy must be stable for 5 days prior to scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)

Hepatic

* SGOT < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* No active or latent hepatitis B infection

Renal

* Creatinine < 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled significant medical illness that would preclude study treatment
* No active infection
* No active HIV infection
* No concurrent disease that would dangerously alter drug metabolism or obscure toxicity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 7 days since prior interferon or thalidomide
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent immunotherapy

Chemotherapy

* No prior temozolomide
* At least 14 days since prior methotrexate
* At least 21 days since prior procarbazine
* At least 42 days since prior nitrosoureas
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 7 days since prior tamoxifen
* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* Recovered from all prior therapy
* At least 28 days since prior investigational agents
* At least 28 days since other prior cytotoxic therapy
* At least 7 days since other prior non-cytotoxic agents (e.g., tretinoin) (radiosenitizers allowed)
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nayak L, Abrey LE, Drappatz J, et al.: Multicenter phase II trial of temozolomide (TMZ) and rituximab (RIT) for recurrent primary CNS lymphoma (PCNSL): North American Brain Tumor Consortium (NABTC) study 05-01. [Abstract] J Clin Oncol 29 (Suppl 15): A-2039, 2011.
- [Derived] Nayak L, Abrey LE, Drappatz J, Gilbert MR, Reardon DA, Wen PY, Prados M, Deangelis LM, Omuro A; North American Brain Tumor Consortium. Multicenter phase II study of rituximab and temozolomide in recurrent primary central nervous system lymphoma. Leuk Lymphoma. 2013 Jan;54(1):58-61. doi: 10.3109/10428194.2012.698736. Epub 2012 Jul 9. PMID 22656234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients enrolled from 2005 through 2008. Patients enrolled in an outpatient multi-institutional clinics
Groups:
- IV Rituximab: IV Rituximab 750mg/m2 single infusion every week for up to 4 weeks.
  Induction: Rituximab (750mg/m2) Day 1, 8, 15 and 22 and Temozolomide [TMZ] (150mg/m2) days 1-7 and 15-21, followed by six cycles of consolidation TMZ 150-200mg/m2 x5/28days, followed by maintenance with methylprednisolone (1g IV every 28days) until progression
  rituximab: given IV days 1,8, 15 and 22
  methylprednisolone: 2hr IV every 28 days post consolidation cycles of Temozolomide (TMZ) (6 cycles TMZ = Consolidation cycles)
  temozolomide: Induction Days 1-7 and 15-21 (150mg/m2 PO) Consolidation days 1-5 every 28 days X 6 cycles
Period: Overall Study
Arm/Group | IV Rituximab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Rituximab
Number analyzed (Participants) | 16
Age, Customized [Median (Full Range); unit: years] | 63 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate of the combination of Rituximab and TMZ
Time Frame: 2 months
Population: 2 patients were not evaluable, one died prematurely and the other withdrew consent before the first scan (during induction cycle)
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | IV Rituximab
Number analyzed (Participants) | 14
percent of participants | 14 [2 to 43]

2. Secondary Outcome: Number of Participants Alive at 3 Years
Description: The intent was to measure Median Overall Survival at 3 years, however only one participant was analyzable at this time point. Therefore, the number of participants who survived is reported instead.
Time Frame: 3 years
Population: One patient died prematurely, one patient withdrew consent before first scan (during induction), 13 patients came off study due to progression of disease.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Rituximab
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: 1 Year Overall Survival Rate
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IV Rituximab
Number analyzed (Participants) | 16
percentage of participants | 71 [40 to 88]

4. Secondary Outcome: 6-month Progression-free Survival
Description: Scan at 6 months
  Complete response: Complete disappearance of all tumor on MRI scan, off all glucocorticoids with stable or improving neurological exam minimum of 4 wks
  Partial response: Greater than or equal 50% reduction in tumor size on MRI, on sable or decreasing glucocorticoids with stable or improving neurological exam for a minimum of 4 wks.
  Progressive disease: Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
  Stable disease: Clinical status and MRI does not qualify for complete response, partial response or progression
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IV Rituximab
Number analyzed (Participants) | 16
percentage of participants | 13 [2 to 35]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | IV Rituximab
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Rituximab (N=16)
fatigue (General disorders) | 3 (3)
liver enzyme elevation (Investigations) | 2 (2)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
hematotoxicity (Blood and lymphatic system disorders) | 8 (8)

LIMITATIONS AND CAVEATS:
slow accrual, preliminary analysis suggesting futility and combining of consortia, trial closed early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No